CLINICAL TRIAL: NCT06420908
Title: Induction Adebrelimab Combined With Chemotherapy Followed by Concurrent Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma (ESCC): A Prospective, Single-arm, Phase II Clinical Study
Brief Title: Adebrelimab Combined With Chemoradiotherapy for Locally Advanced Unresectable Esophageal Squamous Cell Carcinoma (ESCC)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary reason for termination was difficulty in recruitment
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, Principal Investigator, Hebei Medical University Fourth Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARL-ESCC-001
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PET-CT responders (Experimental): SUV (PETr) reduction >35%
  Interventions: Drug: Adebrelimab+TP/FP+ radiation therapy
- PET-CT non-responders (Experimental): SUV (PETr) reduction ≤35%
  Interventions: Drug: Adebrelimab+FP/TP+ radiation therapy

INTERVENTIONS:
Drug: Adebrelimab+TP/FP+ radiation therapy — Induction stage：
  Adebrelimab : 1200mg d1, iv, q3w TP : nab-paclitaxel paclitaxel 180mg/m2, or paclitaxel 135-175mg/m2, d1, iv; carboplatin AUC=5-6, d1, iv, q3w FP : fluorouracil 400mg/m2, 2400 mg/m2 (48 hours), d1; cisplatin 75mg/m2, d1, iv, q3w 2 cycles;
  Treatment stage:
  TP : nab-paclitaxel paclitaxel 60-70mg/m2, or paclitaxel 75mg/m2, d1, iv; carboplatin AUC=5, d1, iv, q3w FP : fluorouracil 300mg/m2/d, iv; cisplatin 75mg/m2, d1, iv, q3w Radiation therapy (50.4Gy-60Gy/28-33f);
  Consolidation stage:
  Adebrelimab: 1200mg d1, iv, q3w , until disease progression or unacceptable toxicity occurs.
  Arms: PET-CT responders
Drug: Adebrelimab+FP/TP+ radiation therapy — Induction stage：
  Adebrelimab : 1200mg d1, iv, q3w TP : nab-paclitaxel paclitaxel 180mg/m2, or paclitaxel 135-175mg/m2, d1, iv; carboplatin AUC=5-6, d1, iv, q3w FP : fluorouracil 400mg/m2, 2400 mg/m2 (48 hours), d1; cisplatin 75mg/m2, d1, iv, q3w 2 cycles;
  Treatment stage: (switch to a different chemotherapy drug which not used during the earlier induction phase)
  FP : fluorouracil 300mg/m2/d, iv; cisplatin 75mg/m2, d1, iv, q3w TP : nab-paclitaxel paclitaxel 60-70mg/m2, or paclitaxel 75mg/m2, d1, iv; carboplatin AUC=5, d1, iv, q3w Radiation therapy (50.4Gy-60Gy/28-33f);
  Consolidation stage:
  Adebrelimab: 1200mg d1, iv, q3w , until disease progression or unacceptable toxicity occurs.
  Arms: PET-CT non-responders

SUMMARY:
This study aims to evaluate the efficacy and safety of induction Adebrelimab (anti-PD-L1 antibody) combined with chemotherapy, then guided by PET-CT assessment to change the following chemoradiotherapy regiment for locally advanced unresectable ESCC.

ELIGIBILITY:
Inclusion Criteria:

1.Age 18-75 years old, both men and women; 2.Histopathology confirmed as esophageal squamous cell carcinoma，stage II-IVa：T1N2-3M0，T2-4bN+M0； 3.If technically feasible, all patients are recommended to have local staging determined by endoscopic ultrasound (EUS); The endoscopic examination report or gastrointestinal (GI) clinical records should clearly indicate the T and N stages; Perform PET-CT examination; 4.Except for basal or squamous cell skin cancer, bladder cancer in situ or cervical cancer, there is no history of malignant tumor within 5 years; Patients with malignant tumors who have undergone surgical treatment in the past and those who have survived disease-free for more than 5 years meet the inclusion criteria; 5.Have not received any systemic anti-tumor treatment in the past (systemic chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.) 6.According to RECIST 1.1, at least one measurable lesion; 7.ECOG: 0~1; 8.Expected survival period ≥ 12 weeks; 9.Major organ function has to meet the following certeria:

1. Blood routine examination:

   1. HB≥90g/L;
   2. ANC ≥ 1.5 × 109 / L;
   3. PLT ≥ 100 × 109 / L;
2. Biochemical examination:

   1. ALT and AST < 2.5×ULN;
   2. TBIL ≤ 1.5×ULN;
   3. Cr ≤ 1.5×ULN; 9. Left ventricular ejection fraction (LVEF) ≥50%; 11. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; negative serum or urine pregnancy test within 7 days prior to study enrollment And must be non-lactating patients; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period; 12. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Previous history of esophageal cancer surgery；
2. Higher risk of esophageal perforation or fistula；
3. Received systemic immunosuppressive therapy within 14 days prior to the first study medication；
4. Known or suspected to have interstitial pneumonia; Other moderate to severe lung diseases that may seriously affect respiratory function;
5. The patient has any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, enteritis, systemic lupus erythematosus, rheumatoid arthritis; patients with vitiligo, Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
6. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 1000 copies/ml or 500IU/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method)；
7. Within 6 months, cerebral vascular accidents (including transient ischemic attacks or symptomatic pulmonary embolism) occur;
8. History of cardiovascular disease with significant clinical significance, including but not limited to: (1) congestive heart failure (NYHA grade>2); (2) Unstable angina pectoris; (3) Have experienced myocardial infarction within 3 months; (4) Any supraventricular arrhythmias or ventricular arrhythmias that require treatment or intervention;
9. Severe infections within 4 weeks before study drug administration, or active infection with CTCAE ≥ 2 grade treated with antibiotics within 2 weeks before study drug administration;
10. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
11. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
12. The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
1. Objective response rate (ORR) | tumor assessment every 6 weeks since the treatment began，up to 24 monthss
  Baseline to measured stable disease
2. Duration of Overall Response（DoR） | tumor assessment every 6 weeks since the treatment began，up to 24 months
  The duration of overall response is measured from the time that measurement criteria are met for complete response or partial response until the first date that recurrent or progressive disease is objectively documented.
3. Overall survival (OS) | the first day of treatment to death or last survival confirm date,up to 24 months
  Baseline to measured date of death from any cause
4. Adverse events | up to 24 months
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. The number of Participants with adverse events will be recorded at each treatment visit.